CLINICAL TRIAL: NCT01099345
Title: A Pilot, Overactive Bladder Syndrome Study Utilizing a Sleep Laboratory Setting to Compare Detrusor Positive Nocturia Female Subjects to Detrusor Negative Nocturia Female Subjects
Brief Title: A Pilot Trial in a Sleep Laboratory Setting to Observe Night Time Bladder Function of Subjects With Overactive Bladder (OAB)
Status: Terminated | Type: Observational
Why Stopped: Slow Enrollment
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 905-UC-040
Record Dates: First submitted 2010-03-30; First posted 2010-04-07 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Bladder Function
Keywords: OAB; Nocturia; Bladder function; cystometry; polysomnography
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 - OAB with DO+: Subjects that DO+ nocturia
  Interventions: Procedure: cystometry (CMG); Procedure: polysomnography (PSG)
- Group 2- OAB with DO-: Subjects that DO- nocturia
  Interventions: Procedure: cystometry (CMG); Procedure: polysomnography (PSG)

INTERVENTIONS:
Procedure: cystometry (CMG) — recording device measuring pressures though catheters placed in bladder and rectum
Procedure: polysomnography (PSG) — Recording device measuring sleep activity through electrodes attached to the subject

SUMMARY:
This is an observational, pilot, non-treatment study to evaluate and develop clinical variables for distinguishing female OAB subjects that have detrusor overactivity positive (DO+) nocturia from female OAB subjects that have detrusor overactivity negative (DO-) nocturia utilizing a sleep laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have confirmed diagnosis of OAB and OAB symptoms for ≥ 3 months
* Subject must have documented detrusor overactivity
* Subject must not be taking any OAB medication for at least 14 days
* Subject has no sleep related conditions (other than nocturia)

Exclusion Criteria:

* Subject has active urinary tract infection (UTI)
* Subject has significant stress incontinence or mixed stress/urge incontinence
* Subject has nocturnal polyuria
* Subject has history of sleep apnea
* Subject has indwelling urinary catheterization within 4 weeks
* Subject using medication that effects urinary and sleep function
* Subject is unable to refrain from alcohol or smoking during the sleep night stay
* Subject has an unstable medical or psychiatric disorder
* Subject has a history of cardiovascular concerns
* Subject is pregnant, breastfeeding or plans to become pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified through urology physicians, family practice physicians and advertising
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Average nocturia individual volume void | During night in sleep lab
Nocturnal functional bladder capacity | During night in sleep lab
Total urine production | During night in sleep lab

SECONDARY OUTCOMES:
Total wake time from lights out until getting out of bed in the morning | During night in sleep lab
Average urgency rating | During night in sleep lab
Number of nocturias with urgency ≥3 | During night in sleep lab
Percentage of subjects with ≥ 2 nocturias | During night in sleep lab
Time from awakening to void on CMG/PSG | During night in sleep lab
Number of awakenings | During night in sleep lab
Wake time after sleep onset | During night in sleep lab
Sleep onset latency | During night in sleep lab
For DO+ subjects, number of nocturias associated with DO+ | During night in sleep lab

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States